CLINICAL TRIAL: NCT00329524
Title: Using PET-CT to Target and Validate Low-frequency TMS as Treatment for Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Tinnitus Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 51817
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Results first posted 2009-08-07 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Tinnitus
Keywords: Tinnitus; TMS; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active versus Sham Treatment (Sham Comparator): Subjects randomly assigned to active and sham TMS separated by one week interval.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — TMS will initially be targeted to asymmetric cortical activation in one hemisphere, as defined by PET-CT imaging. TMS will then be optimized by identifying the area of maximal tinnitus suppression, within the area of asymmetry, by delivering single 1-Hz pulses of TMS at the MT. The area of maximal tinnitus suppression, as reported by the patient, will then be targeted for treatment with rTMS at 1-Hz frequency, delivering 1800 pulses at 110% MT on each of 5 consecutive treatment days.If no area of maximal tinnitus suppression can be found in the hemisphere initially targeted for treatment based on PET, we will perform the optimization procedure in a homologous region of the opposite cerebral hemisphere to determine if a maximal area of suppression can be found there. Each group will then crossover to sham and active stimulation conditions, respectively, 7 days following the completion of the first treatment session.

SUMMARY:
One out of every five people experience tinnitus (a buzzing, ringing, or roaring sound in the ear) ranging from mild to severe impairment. To date there is no effective therapy that seems to help the tinnitus sufferer. The purpose of this study is to develop a therapy using a technique called Repetitive Transcranial Magnetic Stimulation (rTMS) to hopefully alleviate or reduce the symptoms of tinnitus.

This research is being conducted at the University of Arkansas for Medical Sciences (UAMS). Up to twenty (20) right handed subjects, either males or females, 19-65 years of age, with tinnitus that is severe enough for those persons to seek medical attention will have been seen as patients in the UAMS Hearing and Balance Center, where routine testing includes a physical exam, hearing tests, evaluation of middle ear status, and an MRI scan (a machine that acquires visual images of the brain). A diagnosis of tinnitus will be established after ruling out all other possible causes of the tinnitus.

DETAILED DESCRIPTION:
Subjects will be up to 20 right-handed patients (men and women), 19-65 years of age, with debilitating unilateral or bilateral tinnitus. All subjects must report experiencing the presence of their phantom auditory perception for at least 6 months and have a Tinnitus Handicap Questionnaire (THQ) score >30. Subjects will be recruited from the Otolaryngology Clinic at UAMS, where routine testing includes a physical exam; pure tone audiometry; and evaluation of middle ear status using tympanometry, stapedius reflex tests, and otoscopy. Patients will undergo a gadolinium-contrast MRI of the head to rule out acoustic neuroma or any other central nervous system pathology. All subjects will be thoroughly informed of the risks associated with the procedures in this study, as described in the Hazards to Subjects section, and written informed consent will be obtained. Subjects will be recruited for this study without regard to race or ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* right-handed subjects
* 19-65 years of age
* debilitating unilaterial or bilateral tinnitus
* Experiencing the presence of phantom auditory preception for >6 months
* Tinnitus Handicap Questionnaire score of >30

Exclusion Criteria:

* significant neurological disease
* acoustic neuromas or glomus tumors
* active Meniere's disease
* profound hearing loss
* non English speaking
* personal or family history of epilepsy
* personal history of head injury, aneurysm, stroke, previous cranial neurosurgery, neurological or psychiatric disorders, metal implants in the head or neck, a pacemaker, pregnancy, migraines,
* medications that lower seizure threshold and are contraindicated
* individuals who have been taking certain medications
* claustrophobia
* patients who do not exhibit significant cortical asymmetries on PET

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-06; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Dornhoffer, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Result] Smith JA, Mennemeier M, Bartel T, Chelette KC, Kimbrell T, Triggs W, Dornhoffer JL. Repetitive transcranial magnetic stimulation for tinnitus: a pilot study. Laryngoscope. 2007 Mar;117(3):529-34. doi: 10.1097/MLG.0b013e31802f4154. PMID 17334317
- [Result] Richter GT, Mennemeier M, Bartel T, Chelette KC, Kimbrell T, Triggs W, Dornhoffer JL. Repetitive transcranial magnetic stimulation for tinnitus: a case study. Laryngoscope. 2006 Oct;116(10):1867-72. doi: 10.1097/01.mlg.0000234936.82619.69. PMID 17016213

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Versus Sham TMS: Active or sham TMS will initially be targeted to asymmetric cortical activation in one hemisphere, as defined by PET-CT imaging according to a randomized schedule. This area will then be targeted either for active treatment with rTMS at 1-Hz frequency, delivering 1800 pulses at 110% MT on each of 5 consecutive treatment days or sham treatment of the same duration.
Period: Overall Study
Arm/Group | Active Versus Sham TMS
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Active Versus Sham TMS
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in PET Asymmetry Index
Description: Change in calculated PET asymmetry index between left and right temporal lobe from baseline following active Tx
Time Frame: After active treatment week
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Active Versus Sham TMS
Number analyzed (Participants) | 5
ratio | 1.2 (2.3)

2. Secondary Outcome: Psychomotor Vigilance
Description: Change in simple auditory reaction time after treatment
Time Frame: Immediately after treatment
Population: per protocol
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Active Versus Sham TMS
Number analyzed (Participants) | 5
milliseconds | -30 (18.27)
Statistical Analysis 1: Comparison: Active Versus Sham TMS; Test type: Non-Inferiority or Equivalence — Power analysis based on paired t-test; p < .05, t-test, 2 sided

3. Secondary Outcome: Difference in Visual Analog Rating of Tinnitus (VAR)Following Active and Sham Tx
Description: Rating of tinnitus loudness using a scale of 0-100 for
Time Frame: immediately following active and sham TMS
Measure: Mean (Standard Deviation); unit: analog rating
Arm/Group | Active Versus Sham TMS
Number analyzed (Participants) | 5
analog rating | 2.5 (1.2)
Statistical Analysis 1: Comparison: Active Versus Sham TMS; Test type: Superiority or Other; p = .05, test for order effect

ADVERSE EVENTS:
Groups:
- Active Versus Sham Treatment: Subjects randomly assigned to active and sham TMS separated by one week interval.
  Repetitive Transcranial Magnetic Stimulation (rTMS): TMS will initially be targeted to asymmetric cortical activation in one hemisphere, as defined by PET-CT imaging. TMS will then be optimized by identifying the area of maximal tinnitus suppression, within the area of asymmetry, by delivering single 1-Hz pulses of TMS at the MT. The area of maximal tinnitus suppression, as reported by the patient, will then be targeted for treatment with rTMS at 1-Hz frequency, delivering 1800 pulses at 110% MT on each of 5 consecutive treatment days.If no area of maximal tinnitus suppression can be found in the hemisphere initially targeted for treatment based on PET, we will perform the optimization procedure in a homologous region of the opposite cerebral hemisphere to determine if maximal area of suppression can be found there. Each group will then crossover to sham and active stimulation conditions, respectiv
Arm/Group | Active Versus Sham Treatment
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
Study was ended early and analysis was limited to only 5 subjects. A follow up study using a revised protocol is underway.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No